CLINICAL TRIAL: NCT02948725
Title: Clinical Application of Cross-education During Stroke Rehabilitation
Acronym: X-Ed-Stroke01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Jonathan Farthing, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: X-Ed-Stroke01
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cross-education + standard rehabilitation (Experimental): The cross-education group will engage in strength training of the non-paretic hand in addition to standard rehabilitation. Cross-education will be progressive in nature, beginning with 2 sets of 8 repetitions and increasing up to a maximum of 6 sets of 8 repetitions of maximal voluntary effort isometric handgrip contractions as tolerated. Grip training will be performed using standard grip trainers (Digi-Flex Grip trainers) to train both finger flexors and full hand and wrist isometric contractions. In addition, patients will perform controlled dynamic wrist flexion and extension training of the non-paretic hand using exercise tubing with the same prescription. Patients will be asked to complete exercises 3 times per week for 26 weeks, and to record adherence in a training log. An average of one session per week will be considered 'trained'.
  Interventions: Other: Cross-education + standard rehabilitation
- standard rehabilitation (No Intervention): Standardized rehabilitation involves several strategies tailored to the patient and remains somewhat based on clinician preference. These therapies may involve functional electrical stimulation, neuro-facilitation, strengthening, range of motion (ROM), mirror therapy, and force-use therapy (e.g., CIMT). Patients engage in therapy 5 days per week as inpatients, and 2 days per week as outpatients with additional home exercises. Specific therapies for each patient will be tracked using a therapy log.

INTERVENTIONS:
Other: Cross-education + standard rehabilitation
  Arms: cross-education + standard rehabilitation

SUMMARY:
Based on the current state of knowledge and gaps in the literature we will conduct an intervention study to explore novel treatment and rehabilitation of patients at Royal University Hospital (RUH) with motor deficits following stroke. This project has the following objectives:

1. To determine if cross-education, in addition to standard rehabilitation leads to better recovery of upper limb function for stroke patients with hemiparesis.
2. To incorporate functional brain activation as measured by functional magnetic resonance imaging (fMRI) to examine the neural mechanisms associated with changes in motor function of the paretic arm post-stroke.
3. To use diffusion tensor imaging (DTI) tractography to measure connectivity and examine the extent to which white matter tract thickness correlates with preserved motor output in patients post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* within 18 months of stroke recovery
* medically stable
* ambulatory
* have moderate to severe upper limb hemiparesis as diagnosed by clinicians
* Consent

Exclusion Criteria:

* significant cognitive impairment or aphasia affecting understanding, as assessed by clinician
* severe upper limb spasticity preventing any movement of the proximal arm and shoulder
* diagnosis of hemorrhagic or bilateral stroke
* history of other severe upper limb musculoskeletal injury
* other neurological diseases
* intracranial metal clips or cardiac pacemaker, or anything that would preclude an MRI
* Any condition that would preclude the participant's ability to attend follow-up visits in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Motor function scores as assessed using the Fugl-Meyer Assessment | At 26 weeks

SECONDARY OUTCOMES:
grip and wrist strength | At 26 weeks
volume of motor cortex activation | At 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jon Farthing, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Co-Investigators will have access to the data. Plans beyond that